CLINICAL TRIAL: NCT05271721
Title: Trans-foraminal Lumbar Epidural Injection of Dexmedetomidine Against Magnesium Sulfate When Combined With Dexamethasone in Uni-lateral Lower Limb Radicular Pain. Multi-centeric Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R/219
Record Dates: First submitted 2022-02-26; First posted 2022-03-09 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Other): Dexamethasone 4 mg (1ml) plus 40 mg ( 2ml) lidocaine 2% plus 1ml sterile saline
  Interventions: Drug: transforaminal epidural injection of dexamethasone
- Magnesuim group (Active Comparator): . 200 mg Mg sulfate (1ml) plus 4 mg dexamethasone(1ml) plus 40mg lidocaine 2% (2ml)
  Interventions: Drug: epidural transforaminal injection of magnesuim sulfate
- Dexmedetomidine group (Active Comparator): Dexmedetmodine 50mic (0.5ml) ,4 mg dexamethasone (1ml), 40 mg lidocaine 2% (2ml) added to 4ml total volume with sterile saline .
  Interventions: Drug: epidural transforaminal injection of dexmedtemodine

INTERVENTIONS:
Drug: epidural transforaminal injection of magnesuim sulfate — transforaminal fluroscopic guided
  Other Names: floroscopic epidural injection of magnesuim
  Arms: Magnesuim group
Drug: epidural transforaminal injection of dexmedtemodine — transforaminal fluroscopic guided
  Other Names: fluroscopic eoidural injection of dexmedtemodine
  Arms: Dexmedetomidine group
Drug: transforaminal epidural injection of dexamethasone — transforaminal fluroscopic guided
  Other Names: fluroscopic epidural injection of dexamethasone
  Arms: control group

SUMMARY:
Transforaminal injection of chronic radicular lower limb injection by either dexmedetomdine or magnesuim sulfate

ELIGIBILITY:
Inclusion Criteria:

* Age group. 25-75ys old
* Both sex.
* Lumber disc protrusion at one or two segments on MRI.
* Chronic lumbar radiculer pain for more than 6 weeks refractory to
* medical treatment for at least 4 weeks. .
* Positve leg rising test at 30-70 degrees.

Exclusion Criteria:

* Diabetic candidates ( type Ior II).
* Patient refusal.
* MRI with disc sequestration.
* Neurological examination revealed foot drop, neuropathic ulcers
* Myelopathic or scoliotic patients, .
* Coagulopathic patients ( cirrhotic patients, on anti-coagulation )

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
pain score | up to 6 months post-injection
  visual analogue pain score. pain value of (0 cm) equals no pain , and value of (10 cm) equals worst pain

SECONDARY OUTCOMES:
functional disability | up to 6 months post injection
  Modified Oswestry Disability Questionnaire....0% to 20%: minimal disability:....21%-40%: moderate disability: 41%-60%: severe disability...61%-80%: crippled
acute complications | 6 hours post-injection
  number of patients developed epidural hematoma by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Minia University Hospital, Egypt